CLINICAL TRIAL: NCT00902980
Title: Regional Transplant Programs Study of Immunosuppressive Therapy Related Toxicities in Renal Transplant Recipients Managed at Regional or Satellite Community Nephrology Clinics
Brief Title: Study of Immunosuppressive Therapy Toxicities in Kidney Transplant Recipients at Regional or Satellite Community Clinics
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma Canada, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: FKC-010
Record Dates: First submitted 2009-05-13; First posted 2009-05-15 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Kidney Transplantation
Keywords: Kidney transplantation; Tacrolimus; Immunosuppression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1. Community Based Clinics: Patient charts from community based nephrology clinics
  Interventions: Other: Chart Review
- 2. Regional Clinics: Patient charts from regional transplant clinics
  Interventions: Other: Chart Review

INTERVENTIONS:
Other: Chart Review — Chart review of patients / graft outcome in renal transplant recipients

SUMMARY:
This is a multicentre, observational, non-interventional, retrospective analysis by chart review.

DETAILED DESCRIPTION:
This study will compare differences in patient and graft related outcomes in renal transplant recipients followed in regional transplant centers versus satellite clinics.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 months post transplant
* Patient had the current transplant during the period 1 July 1997 to no less than 18 months prior to chart review
* Patient is currently on tacrolimus/MMF or AZA - or cyclosporine/MMF or AZA based immunosuppressive therapy
* Patient is not a recipient of dual kidney or multi -organ transplant
* Patient has a functioning graft (i.e. patient does not require dialysis)
* Patient is recipient of a renal transplant including living or cadaveric, related or non-related, or pediatric en bloc kidneys, but excluding kidney-pancreas transplant recipients
* Patient received the current transplant at one of six identified regional transplant centers
* Patient is currently followed in a regional or satellite community based nephrology clinic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Canadian subjects post renal transplant, currently being treated with immunosuppressive therapy
Sampling Method: Probability Sample
Enrollment: 264 (Actual)
Dates: Start 2005-04; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Change in renal function over 6-18 months estimated by change in serum creatinine and glomerular filtration rate (GFR) | 6, 12 and 18 months

SECONDARY OUTCOMES:
Prevalence of hyperlipidemia, hypertension, weight gain/central adiposity, hypertrichosis, alopecia, diabetes mellitus, bone disease and gingival hyperplasia | 6, 12 and 18 months
Comparison of patients on cyclosporine-vs. tacrolimus-based immunoprophylaxis as well as community-based vs. regional transplant nephrology clinics in both incidence of toxicities and related clinical interventions | 6, 12 and 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Canada, Inc.
Locations (12):
- Canada (12):
  - New Westminster, British Columbia
  - Vancouver, British Columbia
  - Moncton, New Brunswick
  - Saint John, New Brunswick
  - Halifax, Nova Scotia
  - Sydney, Nova Scotia
  - Greater Sudbury, Ontario
  - London, Ontario
  - Mississauga, Ontario
  - Sault Ste. Marie, Ontario
  - Thunder Bay, Ontario
  - Toronto, Ontario

REFERENCES:
- [Background] Keough-Ryan TM, Prasad GV, Hewlett T, Shapiro RJ; Canadian Community Nephrology Study Group. Similar outcomes for Canadian renal transplant recipients followed up in transplant centers and satellite clinics. Transplantation. 2010 Sep 27;90(6):591-6. doi: 10.1097/tp.0b013e3181e9febd. PMID 20865815
- [Background] Prasad GV, Nash MM, Keough-Ryan T, Shapiro RJ. A quality of life comparison in cyclosporine- and tacrolimus-treated renal transplant recipients across Canada. J Nephrol. 2010 May-Jun;23(3):274-81. PMID 20383867